CLINICAL TRIAL: NCT05558930
Title: MRI-navigated Cerebellar Intermittent Theta-Burst Stimulation（iTBS）in Patients With Disorders of Consciousness
Brief Title: Cerebellar iTBS in Patients With Disorders of Consciousness
Acronym: CTPDOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20222028
Record Dates: First submitted 2022-09-01; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-05

CONDITIONS: Disorder of Consciousness; Vegetative State; Minimally Conscious State
Keywords: TMS; cerebellar; iTBS; DOC; MCS; VS
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State

STUDY DESIGN:
Intervention Model Description: A randomized double-blinded, sham-controlled, crossover study design is used to investigate the effects of bilateral cerebellar iTBS on patients with prolonged DOC in a VS/UWS or in a MCS state. We prospectively recruit 44 patients in VS/UWS or MCS state. Each patient will receive bilateral cerebellar iTBS and sham stimulation in random order, one session per day for 5 consecutive days, separated by a 5-day washout. TMS is performed by personalized neuro-navigation to target the cerebellar dentate nucleus. The primary research outcome is whether bilateral cerebellar iTBS, as compared to sham stimulation, will improve consciousness (as measured by changes in CRS-R total scores) in VS/UWS and MCS patients. Secondary research outcome is evaluated by Electroencephalogram(EEG), CRS-R subscore, and Glasgow Outcome Scale-Extended(GOSE) score at 3 and 6 months of enrollment.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iTBS stimulation (Experimental): Participants receive iTBS stimulation of bilateral cerebellar one session per day for 5 consecutive days.
  Interventions: Device: iTBS stimulation
- sham stimulation (Sham Comparator): Participants receive sham stimulation of bilateral cerebellar one session per day for 5 consecutive days.
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: iTBS stimulation — standard iTBS burst pattern:3 pulses at 50-Hz repeated at a rate of 5-Hz; 20 trains of 10 bursts given with 8-s intervals. 600 pulses on both side of cerebellar with an interval of 5 minutes.
  Arms: iTBS stimulation
Device: sham stimulation — Participants receive a sound stimulation with the same pattern with iTBS stimulation,but without magnetic field
  Arms: sham stimulation

SUMMARY:
Previous studies showed the excitatory effect of cerebellar transcranial magnetic stimulation(TMS) on motor cortex.Investigator evaluate the effects of bilateral cerebellar TMS on Coma Recovery Scale-Revised (CRS-R) scores in patients with disorders of consciousness(DOC) in a randomized, double-blinded, sham-controlled, crossover experimental design.

DETAILED DESCRIPTION:
Patients with disorders of consciousness(DOC) resulting from severe brain injury greatly burden caregivers, health care facilities, and society. However, there is no definitively effective treatment for patients with DOC.

Previous studies showed the excitatory effect of cerebellar transcranial magnetic stimulation(TMS) on motor cortex through the dentato-rubro-thalamic tract. Investigators aim to validate the effect of 5 consecutive sessions of intermittent theta-burst stimulation(iTBS) of bilateral cerebellar on level of consciousness of patients in vegetative state(VS)/unresponsive awakening state(UWS)or minimally conscious (MCS) state in a randomized, double-blinded, sham-controlled, crossover study.

TMS is a non-invasive and safe neural regulatory approach that is widely used in depression, schizophrenia, stroke, and Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. VS/UWS or MCS according to diagnostic criteria
2. Age ≥18 years
3. Written informed consent obtained

Exclusion Criteria:

1. Patients in coma
2. Brain injury <1week
3. Presence of metallic hardware in close contact to the discharging coil（such as cochlear implants, or an Internal Pulse Generator or medication pumps）
4. Patients with high risks according to standard questionnaire to screen transcranial magnetic stimulation(TMS) candidates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in CRS-R Total Scores | Baseline and directly after 5 sessions of iTBS and sham stimulation（5 days）
  Whether bilateral cerebellar iTBS would improve consciousness in enrolled patients. CRS-R total score is used to measure level of consciousness of disorder.The coma recovery scale-revised(CRS-R) consists of six subscales addressing auditory, visual, motor, verbal, communication, and arousal functions.The lowest item on each subscale represents reflexive activity and the highest item represents cognitively mediated behavior. Maximum scores of each subscale are summed to obtain the total score (from 0 to 23).The score for each subscale is based on the presence or absence of a specific behavioral response to a sensory stimulus (higher scores are better).

SECONDARY OUTCOMES:
Change in CRS-R Subscale Scores | Baseline and directly after 5 sessions of iTBS and sham stimulation（5 days）
  The coma recovery scale-revised(CRS-R) consists of six subscales addressing auditory, visual, motor, verbal, communication, and arousal functions.The lowest item on each subscale represents reflexive activity and the highest item represents cognitively mediated behavior. The score for each subscale is based on the presence or absence of a specific behavioral response to a sensory stimulus (higher scores are better).
Change of Influence on EEG | Baseline and after 5 sessions of iTBS and sham stimulation（5 days）
  EEG will be monitored on the first and fifth sessions of both iTBS and sham stimulation, from 20 minutes before the start of stimulation until 30 minutes after the end of stimulation.
Influence of time since insult on the results | Participants will be followed for the duration of 0.5 year
  Glasgow Outcome Scale-Extended(GOSE) score will be assessed at 3 and 6 months of enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Air Force Military Medical University, Xi'an, Shaanxi, China